CLINICAL TRIAL: NCT00758953
Title: Pain Associated With Endometriosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lumara Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DZ2-201-601-725036
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Danazol Once Weekly
- 2 (Experimental)
  Interventions: Drug: Danazol Twice Weekly
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo Once Weekly
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo Twice Weekly

INTERVENTIONS:
Drug: Danazol Once Weekly — semi-solid
  Arms: 1
Drug: Danazol Twice Weekly — semi-solid
  Arms: 2
Drug: Placebo Once Weekly — semi-solid
  Arms: 3
Drug: Placebo Twice Weekly — semi-solid
  Arms: 4

SUMMARY:
This study will evaluate the efficacy and safety of an investigational medication compared with placebo in the treatment of pain associated with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Menstruating female 18-50 years of age,
* Regular cycle length of 21 to 35 days with menstrual bleeding that typically lasts no more than 7 days,
* Has pain associated with endometriosis,
* Has a documented history consistent with endometriosis,

Exclusion Criteria:

* Is pregnant or lactating,
* Has a history of or has active thrombosis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2007-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Pain associated with endometriosis | 3 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jim Joffrion, Study Director — Lumara Health, Inc.
Locations (44):
- United States (33):
  - Chandler, Arizona
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Carmichael, California
  - San Diego, California
  - Denver, Colorado
  - Britain, Connecticut
  - West Hartford, Connecticut
  - Aventura, Florida
  - Boynton Beach, Florida
  - Clearwater, Florida
  - Hudson, Florida
  - Tampa, Florida
  - Alpharetta, Georgia
  - Atlanta, Georgia
  - Decatur, Georgia
  - Boise, Idaho
  - Champaign, Illinois
  - Baton Rouge, Louisiana
  - Chesterfield, Missouri
  - Moorestown, New Jersey
  - Winston-Salem, North Carolina
  - Bismarck, North Dakota
  - Fargo, North Dakota
  - Cleveland, Ohio
  - Columbus, Ohio
  - Abington, Pennsylvania
  - West Chester, Pennsylvania
  - Jackson, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Irving, Texas
  - Salt Lake City, Utah
- Canada (9):
  - Kelowna, British Columbia
  - North Vancouver, British Columbia
  - Penicton, British Columbia
  - Halifax, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Whitby, Ontario
  - Windsor, Ontario
  - Saskatoon, Saskatchewan
- Russia (2):
  - Moscow
  - Saint Petersburg